CLINICAL TRIAL: NCT04568655
Title: The Noninvasive Ventilation to COVID-19 Patients With Respiratory Failure
Brief Title: The Noninvasive Ventilation to COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhang Jianheng, The First Affiliated Hospital of Guangzhou Medical University, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: FAHGuangzhouYLS03
Record Dates: First submitted 2020-09-28; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Noninvavie Ventilation to Patients With COVID-19
Keywords: noninvavie ventilation; COVID-19; respiratory failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients need noninvasive ventilation
  Interventions: Device: noninvasive ventilation

INTERVENTIONS:
Device: noninvasive ventilation — noninvasive ventilation to support the COVID-19 patients with respiratory failure

SUMMARY:
Noninvasive ventilation(NIV) is an important treatment to the respiratory failure patients.The severe Corona Virus Disease-19(COVID-19) patients are incline to respiratory failure.The NIV may reduce the intubtion rate.This research was taken to investigate the factor to the success of the noninvasive ventilation to the COVID-19 patients with respiratory failure.

DETAILED DESCRIPTION:
Noninvasive ventilation(NIV) is an important treatment to the respiratory failure patients.The severe Corona Virus Disease-19(COVID-19) patients are incline to respiratory failure.The NIV may reduce the intubtion rate.This research was taken to investigate the factor to the success of the noninvasive ventilation to the COVID-19 patients with respiratory failure.We wish to raise the success rate to COVID-19 patients with respiratory failure.More critically ill COVID-19 patients could avoid the intubtion.

ELIGIBILITY:
Inclusion Criteria:

1. Shortness of breath, RR>30 times per minute;
2. At room air, SpO2 lower than 93%;
3. The partial pressure of Arterial blood oxygen (PaO2)/the fraction of inspired oxygen (FiO2) ≤ 300mmHg;
4. CT（computed tomography） chest imaging shows that lung damage develops significantly within 24 to 48 hours.

Exclusion Criteria:

1. Severe cardiovascular disease,
2. respiratory arrest,
3. cardiovascular instability (hypotension, arrhythmias, myocardial infarction),
4. change in mental status or patients who were uncooperative, high risk of aspiration, viscous or copious
5. secretions,
6. recent facial or gastroesophageal surgery,
7. craniofacial trauma, 8)fixed nasopharyngeal abnormalities,

9）burns, 10) extreme obesity.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: respiratory failure patients with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
success rate | 4 month
  the sucess rate of the noninvasive ventilation
the intubtion rate | 4 month
  the intubtion rate of the COVID-19 patients

SECONDARY OUTCOMES:
blood lymphocyte | 4month
  blood lymphocyte of the COVID-19 patients
B-type natriuretic peptide | 4 month
  blood B-type natriuretic peptide of the COVID-19 patients
Procalcitonin | 4 month
  blood procalcitonin of the COVID-19 patients
Oxygen Saturation | 4 month
  Oxygen Saturation of the COVID-19 patients

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
the IPD are going to share after the paper published.